CLINICAL TRIAL: NCT06865144
Title: Prospective, Randomized, Double- Masked Study to Evaluate the Effect of Rhopressa Versus Placebo on Intraocular Pressure (IOP) in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension Post-Selective Laser Trabeculoplasty (SLT)
Brief Title: Effect of Rhopressa on Intraocular Pressure (IOP) in Patients With Primary Open-Angle Glaucoma or Ocular Hypertension Post-SLT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: East Coast Institute for Research (Network)
Collaborators: Alcon, a Novartis Company (Industry); Florida Eye Specialists (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECIR-Alcon-02
Record Dates: First submitted 2025-03-04; First posted 2025-03-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Primary Open Angle Glaucoma or Ocular Hypertension
Keywords: primary open angle glaucoma; ocular hypertension; SLT; POAG; Selective Laser Trabeculoplasty; Rhopressa; netarsudil
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rhopressa (Experimental)
  Interventions: Drug: Netarsudil ophthalmic solution 0.02%
- Artificial Tears (Placebo Comparator)
  Interventions: Drug: Artificial tears

INTERVENTIONS:
Drug: Netarsudil ophthalmic solution 0.02% — Apply one drop in each eye every evening
  Other Names: Rhopressa
  Arms: Rhopressa
Drug: Artificial tears — Apply one drop in each eye every evening
  Arms: Artificial Tears

SUMMARY:
The purpose of this study is to collect data about how Rhopressa affects IOP in patients who have had an SLT procedure in both eyes.

DETAILED DESCRIPTION:
This is a prospective, randomized, double-masked, placebo controlled (artificial tears), single center study. The study population will include seventy (n=70) subjects with POAG or ocular hypertension who have undergone SLT and may benefit from additional IOP reduction. If individuals are a candidate for treatment with Rhopressa (netarsudil) 0.02% ophthalmic solution post-SLT, they can potentially be included in the trial. The study duration per subject is expected to be 6 weeks (or up to 12 weeks if washout is required for previous IOP lowering treatment) with three scheduled study visits.

While both Rhopressa and 360 degrees SLT primarily target the trabecular meshwork, potential synergistic effects of the two therapies on conventional aqueous outflow are not completely understood. This study will determine whether initiation of Rhopressa post-360 degrees SLT provides greater IOP reduction than 360 degrees SLT alone. This information will aid healthcare providers in selecting the best approach to management of IOP in patients who have recently undergone 360 degrees SLT and may benefit from additional IOP reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Documented diagnosis of bilateral POAG or ocular hypertension as determined by the investigator based on medical record review.
3. At Screening (V1), the subject completed SLT in both the eyes within the last 90 days.
4. Mean diurnal IOP of 16 to 28 mmHg at Randomization (V2 )
5. At Randomization (V2), in the opinion of the investigator, subject may benefit from additional IOP reduction in the study eye and is a candidate for treatment with Rhopressa
6. At Randomization (V2), if treated with IOP-lowering medication(s) in either eye prior to SLT, subject has completed the minimum washout period for the medication(s) (see Table 1)
7. If female, subject is either incapable of pregnancy (e.g., history of bilateral oophorectomy, hysterectomy, bilateral tubal ligation) or post-menopausal (amenorrheic for at least 2 years) or will use an effective (e.g., double barrier) method of birth control for the duration of the study

Exclusion Criteria:

1. History of more than one treatment with SLT in either eye
2. Unable or unwilling to discontinue current IOP-lowering medication(s), if applicable
3. Prior or current treatment with a rho kinase inhibitor
4. Prior microinvasive glaucoma surgery (MIGS)
5. Advanced stage of glaucoma, as determined by the investigator based on medical record review
6. Any condition that prevents reliable applanation tonometry in either eye (e.g., significant corneal surface abnormalities, scars, keratoconus)
7. Previous or currently active corneal disease that, in the opinion of the investigator, could affect the study outcomes
8. Active or recurrent intraocular infection, inflammation, iritis or uveitis
9. Retinal disease (e.g., diabetic retinopathy, macular degeneration, central retinal vein or artery occlusion, macular edema)
10. Intraocular injection performed ≤ 6 months prior to Screening (V1)
11. Anticipated use of any topical ocular steroids and/or topical ocular nonsteroidal anti-inflammatory drugs (NSAID) during the study period
12. Current participation in any drug or device clinical investigation, receipt of investigational drug within 6 drug half-lives of Screening (V1), or any previous placement of an investigational device.
13. Any condition in the opinion of the investigator that would potentially confound the results of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Mean diurnal intraocular pressure (IOP) | 42 Days
  Between-group difference in change in mean diurnal IOP

OTHER OUTCOMES:
Intraocular pressure (IOP) reduction at 8am, 10am, and 4pm | 42 Days
  Between-group difference in change in IOP at the 8am, 10am, and 4pm timepoints

CONTACTS AND LOCATIONS:
Locations (1):
- East Coast Institute for Research at Florida Eye Specialists, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP
Time Frame: When the trial starts until it ends data collection

REFERENCES:
- [Background] Stuart, Annie. "Drug Update: Vyzulta and Rhopressa." Glaucoma Clinical Update, 31 Aug. 2018.
- [Background] Zaman F, Gieser SC, Schwartz GF, Swan C, Williams JM. A multicenter, open-label study of netarsudil for the reduction of elevated intraocular pressure in patients with open-angle glaucoma or ocular hypertension in a real-world setting. Curr Med Res Opin. 2021 Jun;37(6):1011-1020. doi: 10.1080/03007995.2021.1901222. Epub 2021 Mar 27. PMID 33733980
- [Background] Gazzard G, Konstantakopoulou E, Garway-Heath D, Garg A, Vickerstaff V, Hunter R, Ambler G, Bunce C, Wormald R, Nathwani N, Barton K, Rubin G, Buszewicz M; LiGHT Trial Study Group. Selective laser trabeculoplasty versus eye drops for first-line treatment of ocular hypertension and glaucoma (LiGHT): a multicentre randomised controlled trial. Lancet. 2019 Apr 13;393(10180):1505-1516. doi: 10.1016/S0140-6736(18)32213-X. Epub 2019 Mar 9. PMID 30862377
- [Background] Kass MA, Heuer DK, Higginbotham EJ, Johnson CA, Keltner JL, Miller JP, Parrish RK 2nd, Wilson MR, Gordon MO. The Ocular Hypertension Treatment Study: a randomized trial determines that topical ocular hypotensive medication delays or prevents the onset of primary open-angle glaucoma. Arch Ophthalmol. 2002 Jun;120(6):701-13; discussion 829-30. doi: 10.1001/archopht.120.6.701. PMID 12049574
- [Background] Allison K, Patel D, Alabi O. Epidemiology of Glaucoma: The Past, Present, and Predictions for the Future. Cureus. 2020 Nov 24;12(11):e11686. doi: 10.7759/cureus.11686. PMID 33391921